CLINICAL TRIAL: NCT01467934
Title: FeverText: Assessing Fever Rates After Influenza and Pneumococcal Vaccination During the 2011-12 Influenza Season Using Text Messaging
Brief Title: FeverText: Assessing Fever Rates After Vaccination During the 2011-12 Influenza Season Using Text Messaging
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Stockwell, MD, MPH, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Other Study IDs: AAAJ0504
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Fever
MeSH Terms: conditions — Fever

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Trivalent inactivated influenza vaccine: Trivalent inactivated influenza vaccine (TIV) 0.25 ml IM x 1
- TIV and PCV13 together: Trivalent inactivated influenza vaccine (TIV) 0.25 ml IM x 1; 13-valent pneumococcal conjugate vaccine (PCV13) 0.5 mL IM x1
- 13-valent pneumococcal conjugate vaccine: 13-valent pneumococcal conjugate vaccine (PCV13) 0.5 mL IM x1

SUMMARY:
In this study, the investigators will prospectively assess fever rates and other associated vaccine adverse events in 6-23 month old patients during days 0-7 after administration of trivalent inactivated influenza vaccine (TIV) and 13-valent pneumococcal conjugate vaccine (PCV13) concomitantly compared to those who receive trivalent inactivated influenza vaccine (TIV) or 13-valent pneumococcal conjugate vaccine (PCV13) administered non-concomitantly. The investigators hypothesize that fever rates will be significantly higher during the 0-1 days after vaccination when inactivated influenza vaccine (TIV) and 13-valent pneumococcal conjugate vaccine (PCV13) are given concomitantly than when TIV or PCV13 is administered non-concomitantly.

ELIGIBILITY:
Inclusion Criteria:

1. are 6 through 23 month olds,
2. have a visit at a study site during the study period of Nov. 1, 2011 through March 31, 2012,
3. receive trivalent inactivated influenza vaccine (TIV)/13-valent pneumococcal conjugate vaccine (PCV13)concomitantly, trivalent inactivated influenza vaccine (TIV)/without 13-valent pneumococcal conjugate vaccine (PCV13) or 13-valent pneumococcal conjugate vaccine (PCV13) without trivalent inactivated influenza vaccine (TIV)/(4) parent has a cell phone with text messaging capabilities; and

(5) parent speaks English or Spanish.

Exclusion criteria:

1. presence of fever >=100.4 at time of vaccination;
2. administration of any antipyretic in the 6-hour period prior to vaccination
3. stated intent to use prophylactic antipyretics at time of vaccination before the development of a fever;
4. stated intention to move away from the NYC area <6 month;
5. parent only speaks a language other than English or Spanish;
6. inability to read text messages;
7. children who received live attenuated influenza vaccine (LAIV) this visit;
8. children who received trivalent inactivated influenza vaccine (TIV) or 13-valent pneumococcal conjugate vaccine (PCV13) in the seven days prior to enrollment date

Note: Patient may receive other vaccines in addition to trivalent inactivated influenza vaccine (TIV)/13-valent pneumococcal conjugate vaccine (PCV13)

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 6-23 months old visiting study sites
Sampling Method: Non-Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Philip LaRussa, MD, Principal Investigator — Columbia University; Karen Broder, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Stockwell MS, Broder K, LaRussa P, Lewis P, Fernandez N, Sharma D, Barrett A, Sosa J, Vellozzi C. Risk of fever after pediatric trivalent inactivated influenza vaccine and 13-valent pneumococcal conjugate vaccine. JAMA Pediatr. 2014 Mar;168(3):211-9. doi: 10.1001/jamapediatrics.2013.4469. PMID 24395025

RESULTS

PARTICIPANT FLOW:
Groups:
- Trivalent Inactivated Influenza Vaccine (TIV) Alone: Trivalent inactivated influenza vaccine 0.25ml IM X 1
- 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone: 13-valent pneumococcal conjugate vaccine (PCV13) 0.5ml IM x 1
Period: Overall Study
Arm/Group | Trivalent Inactivated Influenza Vaccine (TIV) Alone | TIV and PCV13 Together | 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone
Started | 208 | 212 | 110
Completed | 208 | 212 | 110
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Trivalent Inactivated Influenza Vaccine (TIV) Alone: Trivalent inactivated influenza vaccine (TIV) 0.25 ml IM x 1
- 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone: 13-valent pneumococcal conjugate vaccine (PCV13) 0.5 mL IM x1
- Total: Total of all reporting groups
Arm/Group | Trivalent Inactivated Influenza Vaccine (TIV) Alone | TIV and PCV13 Together | 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone | Total
Number analyzed (Participants) | 208 | 212 | 110 | 530
Age, Customized [Number; unit: participants]
  6-11 months | 124 | 145 | 18 | 287
  12-23 months | 84 | 67 | 92 | 243
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 98 | 64 | 263
  Male | 107 | 114 | 46 | 267
Race/Ethnicity, Customized [Number; unit: participants]
  Latino | 171 | 187 | 100 | 458
  Black Latino | 30 | 21 | 9 | 60
  White non-Latino | 4 | 2 | 1 | 7
  Other non-Latino | 3 | 2 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Fever >= 100.4
Time Frame: 8 days
Population: Participants in analysis included those for whom both day 0 and day 1 temperature data was reported.
Measure: Number; unit: percentage of participants
Arm/Group | Trivalent Inactivated Influenza Vaccine (TIV) Alone | TIV and PCV13 Together | 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone
Number analyzed (Participants) | 159 | 170 | 84
percentage of participants | 7.5 | 37.6 | 9.5

ADVERSE EVENTS:
Time Frame: 7 days
Description: medical record review
Arm/Group | Trivalent Inactivated Influenza Vaccine (TIV) Alone | TIV and PCV13 Together | 13-valent Pneumococcal Conjugate Vaccine (PCV13) Alone
Serious Adverse Events (participants affected / at risk) | 0/208 | 0/212 | 0/110
Other Adverse Events (participants affected / at risk) | 0/208 | 0/212 | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No